CLINICAL TRIAL: NCT02920099
Title: Adaptation and Validation of a Nutrition Literacy Assessment Instrument
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 13805; R03HD081730 (NIH)
Record Dates: First submitted 2016-09-27; First posted 2016-09-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Dietary Habits
Keywords: Nutrition literacy
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nutrition Literacy: Participants will be asked to completed the Nutrition Literacy Assessment Instrument (NLAI).
  Interventions: Other: Nutrition Literacy Assessment Instrument (NLAI)

INTERVENTIONS:
Other: Nutrition Literacy Assessment Instrument (NLAI) — Assessment tool which combines elements of different nutrition literacy tools.

SUMMARY:
The purpose of this study is to develop a tool to help researchers better understand what diet information people know and what skills they use to make diet choices.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and read English
* Have 1 or more of the following diseases: diabetes, hyperlipidemia, hypertension, and/or overweight/obesity

Exclusion Criteria:

* Visual acuity insufficient to read the testing instrument
* Cognitive impairment
* Weight > 500 pounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: University of Kansas Medical Center (KUMC) students
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2013-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in Nutrition Literacy Assessment Instrument (NLAI) responses | 1 month
  Participants will complete the NLAI two times over the course of one month. Responses will help shape adaptions to the tool for use in a primary care population.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Gibbs, PhD, RD, LD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States